CLINICAL TRIAL: NCT05308004
Title: Palliative Care Consultations for Persons With Alzheimer's Disease and Related Dementia and Cognitive Impairment in the Medicare Skilled Nursing Facility (SNF) Setting
Brief Title: Palliative Care for Persons With ADRD and CI in SNF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Joan Carpenter, Principal Investigator, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HP-00100348; 3K23NR017663-02S1 (NIH); 1K23NR017663-01A1 (NIH)
Record Dates: First submitted 2022-03-24; First posted 2022-04-01 (Actual); Results first posted 2024-08-14 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Advance Care Planning; Palliative Care; Skilled Nursing Facility; Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Pre-post design where control data will be collected prior to intervention being implemented
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Participants will receive the standard Medicare Skilled Nursing Facility care.
- Palliative Care Consult (Experimental): Participants will receive the standard Medicare Skilled Nursing Facility care plus a Palliative Care Consultation with a trained provider.
  Interventions: Other: Palliative Care Consultation

INTERVENTIONS:
Other: Palliative Care Consultation — Trained provider will discuss illness trajectories, establish and communicate patient-directed goals that guide health care decisions, identify and treat illness-related symptoms, and identify psycho-spiritual needs and approaches to mitigate suffering
  Arms: Palliative Care Consult

SUMMARY:
Alzheimer's disease and related dementias (ADRD) are serious, life limiting illnesses with no known cure. Dementia is the fifth-leading cause of death in older adults and the majority of people with advanced dementia die in nursing homes (NHs). Miller et al reported that 40% of U.S. NH residents dying with advanced dementia received Skilled Nursing Facility (SNF) care in the last 90 days of life, and receipt of this care was associated significantly with poorer end-of-life outcomes, including a higher risk of dying in a hospital, compared to decedents with no SNF care. SNF care is a Medicare post-acute rehabilitation service delivered in NHs focused on intense rehabilitation and/or aggressive, disease-modifying therapies. Regardless of life expectancy, use of SNF care precludes access to Hospice services. Palliative care (PC) offers an evidence-based alternative.

DETAILED DESCRIPTION:
In this pragmatic clinical trial, broadcast notification will be utilized to inform all newly admitted patients at each study site of their participation in this trial. During the admission process, potential subjects will be provided with a 1-page summary sheet (Broadcast notification) detailing their participation in this study that will include contact information for the study team, should the subject or their LAR/surrogate decision maker elect to opt-out of participating.

Baseline data will be collected virtually via telephone by asking each subject or if unable to respond their surrogate decision maker to complete the Patient Outcomes Scale (POSv2), the Satisfaction With Care at the End of Life in Dementia (SWC-EOLD), and the Symptom Management at the End of Life in Dementia (SM-EOLD).

Between 14 days and 21 days after the baseline POSv2, SW-EOLD, and the SM-EOLD are administered, all subjects or if unable to respond their surrogate decision maker will be asked to complete the POSv2, SW-EOLD, and the SM-EOLD again virtually via telephone. The POSv2, SW-EOLD, and the SM-EOLD will be given a total of two times to those in the INTERVENTION and CONTROL groups; at baseline and follow up (14-21 days later).

Deidentified subject demographics will be collected on all participants in the following way: Study team members will review subject's medical records and enter de-identified data into a Research Electronic Data Capture (REDCap) database (Acts staff assists with the study team's access to subject's medical record).

Palliative Care Encounter Trained provider will discuss illness trajectories, establish and communicate patient-directed goals that guide health care decisions, identify and treat illness-related symptoms, and identify psycho-spiritual needs and approaches to mitigate suffering.

ELIGIBILITY:
KEY INCLUSION CRITERIA

Patients:

* Admitted for SNF post-acute care at a participating NHs following a recent hospitalization
* Age ≥ 60 years old
* Speaks English (if verbal)
* If non-verbal/unable to participate in a conversation and/or unable to make decisions, a legally authorized representative (LAR)/surrogate decision maker who can make decisions for the patient as determined by ACTs staff
* Documented ADRD diagnosis in the medical record or history of cognitive impairment (defined as BIMS score ≤ 12)
* At least one global indicator for PC at SNF admission (provider would not be surprised if patient died within 1 year, believes the patient would benefit from advance care planning or symptom management; frequent hospital or NH SNF admissions; complex care requirements; decline in function; feeding intolerance; unintended decline in weight; or previous hospice assessment or enrollment and subsequent discharge)

Surrogate/LAR:

* ≥18 years old
* Family member or friend of an eligible patient as determined by ACTs staff
* Speaks English

KEY EXCLUSION CRITERIA

Patients:

* Who have previously received or are referred for PC by their primary care team
* With a discharge plan within 48 hours of screening
* Currently receiving hospice care
* Who do not have one global indicator of need
* No documented ADRD diagnosis or history of cognitive impairment in the medical record
* That are non-English speaking, (if verbal)
* If unable to make decisions, do not have an LAR/surrogate decision maker.

Surrogate/LAR:

* < 18 years of age
* Not a family Member or friend of an eligible patient
* Non-English speaking

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Acts Continuing Care Retirement Communities, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants enrolled are patients only, not caregivers.
Groups:
- Standard Care: Participants received the standard Medicare Skilled Nursing Facility care.
- Palliative Care Consult: Participants received the standard Medicare Skilled Nursing Facility care plus a Palliative Care Consultation with a trained provider.
Period: Overall Study
Arm/Group | Standard Care | Palliative Care Consult
Started | 4 | 3
Completed | 4 | 2
Not Completed | 0 | 1
Not completed — Not seen by Palliative Care NP | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics were not collected for caregiver participants because they were not enrolled into the study.
Groups:
- Standard Care: Participants (patients) received the standard Medicare Skilled Nursing Facility care.
- Palliative Care Consult: Participants (patients) received the standard Medicare Skilled Nursing Facility care plus a Palliative Care Consultation with a trained provider.
- Total: Total of all reporting groups
Arm/Group | Standard Care | Palliative Care Consult | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 4 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Completed Patient Quality of Life Survey
Description: 12-item survey that measures quality of life in five dimensions: 1) physical; 2) emotional; 3) psychological; 4) spiritual needs, and 5) provision of information and support. Items scored on a 5 point Likert Scale (0=not at all, 4= overwhelmingly) based on symptom/need in the past week. Overall profile score is calculated by summing responses (range 0-40). Source: patient or family caregiver; Time to complete: 5-7 minutes
Time Frame: Collected upon admission to the nursing home (Baseline) and again 21 days post-admission to the nursing home (Follow up)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Palliative Care Consult
Number analyzed (Participants) | 4 | 3
Participants
  Baseline | 4 | 3
  Follow up | 3 | 3

2. Secondary Outcome: Number of Participants That Completed Satisfaction With Care Survey (SWC-EOLD)
Description: 10-item scale that measures caregiver satisfaction with care for persons with dementia. Each item is measured on a 4-point Likert scale ranging from 1 ("strongly disagree") to 4 ("strongly agree"). Specific elements include satisfaction with medical and nursing care, decision-making, and their understanding of the persons with dementia illness. All items are summed, yielding a range of scores of 10-40. Higher scores indicate greater satisfaction.
Time Frame: Collected upon admission to the nursing home and again 21 days post-admission to the nursing home
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Palliative Care Consult
Number analyzed (Participants) | 4 | 3
Participants
  Baseline SWC-EOLD | 4 | 3
  Follow-up SWC-EOLD | 3 | 3

3. Secondary Outcome: Number of Participants That Completed the Symptom Management Survey (SM-EOLD)
Description: 9-item scale administered to a caregiver that measures persons with dementia physical and psychological symptoms. Each item is rated on a 6-point Likert scale ranging from 0 to 5 (0 = "daily", 1 = "several days a week", 2 = "once per week", 3 = "2 or 3 days a month", 4 = "once a month", 5 = "never"). Scores are summed and range from 0 to 45. Higher scores indicate better symptom management.
Time Frame: Collected upon admission to the nursing home and again 21 days post-admission to the nursing home
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Palliative Care Consult
Number analyzed (Participants) | 4 | 3
Participants
  Baseline SM-EOLD | 4 | 3
  Follow-up SM-EOLD | 3 | 3

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Arm/Group | Standard Care | Palliative Care Consult
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT05308004/Prot_SAP_000.pdf